CLINICAL TRIAL: NCT03531242
Title: Phase 2 Open-Label Safety and Immunogenicity Study of the Venezuelan Equine Encephalomyelitis (VEE) Vaccine, Inactivated, Dried, C-84, TSI-GSD 205, Lot 7, Run 1, as Booster Vaccination in Adult Subjects at Risk of Exposure to VEE Virus
Brief Title: Safety and Immunogenicity Study of Venezuelan Equine Encephalomyelitis (VEE) Vaccine as Booster Vaccine in Adults
Acronym: VEE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-13-05
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Venezuelan Equine Encephalomyelitis
MeSH Terms: conditions — Encephalomyelitis, Venezuelan Equine | interventions — Desiccation

STUDY DESIGN:
Intervention Model Description: Subjects who successfully complete screening will be enrolled in the study to receive either (1) a series of booster(s) or (2) one booster vaccination(s). Each vaccination will be administered as 0.5 mL subcutaneous doses in the upper outer aspect of the arm (triceps areas)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Initial Non-responders to VEE TC-83 vaccinations (Experimental): Venezuelan Equine Encephalomyelitis (VEE) Vaccine, Inactivated, Dried, C-84, TSI-GSD 205, Lot 7, Run 1, to be administered as dose(s) of 0.5 mL given subcutaneously in the upper outer aspect of the triceps area.
  Interventions: Biological: 0.5 mL Inactivated, Dried, C-84, TSI-GSD 205, Lot 7, Run 1
- Cohort B: Responders to TC-83 or previous C-84 vaccinations (Experimental): Subjects who showed an initial immune response ≥ 1:20 to TC-83 and whose titer decreased over time or who rollover from a previous VEE C-84 protocol will receive a single 0.5 mL booster dose of C-84 vaccine.
  Subjects who were initial non-responders (< 1:20) to TC-83 will be given subcutaneous 0.5 mL injections on Days 0, 28-35, and 56-63
  Interventions: Biological: 0.5 mL Inactivated, Dried, C-84, TSI-GSD 205, Lot 7, Run 1

INTERVENTIONS:
Biological: 0.5 mL Inactivated, Dried, C-84, TSI-GSD 205, Lot 7, Run 1 — administered as dose(s) of 0.5 mL given subcutaneously in the upper outer aspect of the triceps area. Subjects who showed an initial immune response ≥ 1:20 to TC-83 and whose titer decreased over time or who rollover from a previous VEE C-84 protocol will receive a single 0.5 mL booster dose of C-84 vaccine.
  Subjects who were initial non-responders (< 1:20) to TC-83 will be given subcutaneous 0.5 mL injections on Days 0, 28-35, and 56-63

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of VEE vaccine, C-84, TSI-GSD 205, Lot 7, Run 1, and collect data on the incidence of occupational VEE infection in vaccinated personnel.

DETAILED DESCRIPTION:
Venezuelan Equine Encephalomyelitis Vaccine, Inactivated, Dried, C-84, TSI-GSD 205, Lot 7, Run 1, to be administered as dose(s) of 0.5 mL given subcutaneously in the upper outer aspect of the triceps area. Subjects who showed an initial immune response ≥ 1:20 to TC-83 and whose titer decreased over time or who rollover from a previous VEE C-84 protocol will receive a single 0.5 mL booster dose of C-84 vaccine. Subjects who were initial non-responders (< 1:20) to TC-83 will be given subcutaneous 0.5 mL injections on Days 0, 28-35, and 56-63.

Duration of participation is 12-15 months if the subject demonstrates a PRNT80 of ≥1:20 at 1 year; if not, the vaccination procedure with C-84 will be repeated with a minimum of 28 days between doses. A maximum of four booster doses will be given in a year. If the PRNT80 titer is < 1:20 after four booster doses in any 12-month period, the subject's participation in the study will be placed on hold for 12 months; titers will be repeated at 1 year (± 30 days), and, if required, the subject will be given a booster dose of C-84 vaccine.

Safety endpoint measurements will be evaluated for all subjects receiving at least one vaccination under this protocol regardless of compliance with the protocol. Immunogenicity endpoints will be evaluated for subjects who have been vaccinated in compliance with the protocol and who have had blood for titers drawn in compliance with the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 to 65 years old at time of consent
* Have received VEE TC-83 vaccine
* Have VEE plaque reduction neutralization 80% titers (PRNT80) <1:20
* If female of childbearing potential, must agree to have a urine pregnancy test on the same day before each vaccination administration. (Exception: documented hysterectomy or >3 years of menopause). The results must be negative. Females just agree not to become pregnant for 3 months after receipt of the last study treatment (vaccination).
* Be considered at risk for exposure to VEE virus and who have submitted a Request for IND Vaccines for VDD vaccine.
* Sign and date the approved informed consent document and HIPAA Authorization.
* Have in their charts:
* medical history (including concomitant medications) within 60 days of planned first administration of vaccine
* physical examination and laboratory tests within 1 year
* previous chest radiograph results and electrocardiogram
* Be medically cleared for participation by an investigator (Examinations and/or tests may be repeated at the discretion of the PI).
* Be willing to return for all follow-up visits.
* Agree to report any adverse events (AEs) that may or may not be associated with administration of the vaccine for at least 28 days after administration and agree to report all serious adverse events (for example, resulting in hospitalization) for the duration of the subject's participation in the study.
* Agree to defer blood donation for 1 year after receipt of the vaccine.

Exclusion Criteria:

* Have completed previous VEE C-84 vaccine study as a non-responder.
* Have clinically significant abnormal laboratory results (including evidence of hepatitis C, hepatitis B carrier state) or elevated liver function tests (two times the normal range or at the discretion of the PI).
* Have a personal history of an immunodeficiency or received treatment with an immunosuppressive medication, such as systemically administered glucocorticoids (eg, prednisone) within 1 month before planned administration of the vaccine or with other immunosuppressive therapies within 6 months of planned administration of the vaccine. Other immunosuppressive therapies include all cancer chemotherapeutic agents, drugs to prevent transplant rejection, interferons, monoclonal antibodies, protein kinase inhibitors, methotrexate, TNF (tumor necrosis factor) inhibitors, and any other drug determined to be immunosuppressive by the PI. Current administration of topical, inhalational, or intranasal glucocorticoids is not excluded.
* Have confirmed HIV infection.
* Have positive pregnancy test or be a breastfeeding female.
* Have any known allergies to components of the vaccine:
* Neomycin sulfate
* Streptomycin
* VEE virus, inactivated
* Formaldehyde
* Eggs
* Human serum albumin
* Guinea pig heart cells
* Sodium bisulfite
* Have had a previous serious allergic reaction to guinea pigs or guinea pig products. (Subjects who have known allergies to guinea pigs but whose allergic reactions were not severe may still participate in the study but should be referred to an allergy specialist for assessment and recommendation prior to vaccination).
* Have received or plan to receive another vaccine or investigational product within 28 days of VEE vaccination.
* Have any unresolved AE resulting from a previous immunization.
* Have a medical condition that, in the judgment of the PI, would impact subject safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects Who Develop titers of >1:20 | Month 12-15
  The primary immunogenicity endpoint measurements will be the percentage of per-protocol subjects who develop titers of ≥ 1:20 as determined by PRNT80 after VEE vaccination at each scheduled time point for which blood samples are drawn and over the entire study period to study completion.

SECONDARY OUTCOMES:
GMT for PRNT80 Titers of Subjects at Each Scheduled Time Point | Month 12-15
  The geometric mean PRNT80 titers of per-protocol subjects at each scheduled time point for which blood samples are drawn and over the entire study period to study completion.
Percentage of Subjects with Adverse Events (AEs) Following Vaccination | Month 12-15
  Safety will be evaluated by the nature (body system affected), type [local or systemic], severity, relationship to vaccine, treatment or intervention offered if any, and resolution or outcome) and frequency of AEs for the assessment population
Percentage of Subjects with Each AE Type (local or systemic) | Month 12-15
  Safety will be evaluated by the nature (body system affected), type [local or systemic], severity, relationship to vaccine, treatment or intervention offered if any, and resolution or outcome) and frequency of AEs for the assessment population

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Cardile, DO, MAJ, Principal Investigator — USAMRIID
Locations (1):
- Special Immunizations Program/USAMRIID, Fort Deterick, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossi AL. Rural epidemic encephalitis in Venezuela caused by a group A arbovirus (VEE). Prog Med Virol. 1967;9:176-203. No abstract available. PMID 4383416
- [Background] Casals J, Curnen EC, Thomas L. VENEZUELAN EQUINE ENCEPHALOMYELITIS IN MAN. J Exp Med. 1943 Jun 1;77(6):521-30. doi: 10.1084/jem.77.6.521. PMID 19871301
- [Background] Centers for Disease Control and Prevention (CDC). Venezuelan equine encephalitis--Colombia, 1995. MMWR Morb Mortal Wkly Rep. 1995 Oct 6;44(39):721-4. PMID 7565549
- [Background] Edelman R, Ascher MS, Oster CN, Ramsburg HH, Cole FE, Eddy GA. Evaluation in humans of a new, inactivated vaccine for Venezuelan equine encephalitis virus (C-84). J Infect Dis. 1979 Nov;140(5):708-15. doi: 10.1093/infdis/140.5.708. PMID 528788
- [Background] Franck PT, Johnson KM. An outbreak of Venezuelan encephalitis in man in the Panama Canal Zone. Am J Trop Med Hyg. 1970 Sep;19(5):860-5. doi: 10.4269/ajtmh.1970.19.860. No abstract available. PMID 5453912
- [Background] Hinman AR, McGowan JE Jr, Henderson BE. Venezuelan equine encephalomyelitis: surveys of human illness during an epizootic in Guatemala and El Salvador. Am J Epidemiol. 1971 Feb;93(2):130-6. doi: 10.1093/oxfordjournals.aje.a121233. No abstract available. PMID 5101138
- [Background] Johnson KM, Martin DH. Venezuelan equine encephalitis. Adv Vet Sci Comp Med. 1974;18(0):79-116. No abstract available. PMID 4609399
- [Background] Pittman PR, Makuch RS, Mangiafico JA, Cannon TL, Gibbs PH, Peters CJ. Long-term duration of detectable neutralizing antibodies after administration of live-attenuated VEE vaccine and following booster vaccination with inactivated VEE vaccine. Vaccine. 1996 Mar;14(4):337-43. doi: 10.1016/0264-410x(95)00168-z. PMID 8744562
- [Background] Rivas F, Diaz LA, Cardenas VM, Daza E, Bruzon L, Alcala A, De la Hoz O, Caceres FM, Aristizabal G, Martinez JW, Revelo D, De la Hoz F, Boshell J, Camacho T, Calderon L, Olano VA, Villarreal LI, Roselli D, Alvarez G, Ludwig G, Tsai T. Epidemic Venezuelan equine encephalitis in La Guajira, Colombia, 1995. J Infect Dis. 1997 Apr;175(4):828-32. doi: 10.1086/513978. PMID 9086137
- [Background] SANMARTIN-BARBERI C, GROOT H, OSORNO-MESA E. Human epidemic in Colombia caused by the Venezuelan equine encephalomyelitis virus. Am J Trop Med Hyg. 1954 Mar;3(2):283-93. doi: 10.4269/ajtmh.1954.3.283. No abstract available. PMID 13138831
- [Background] Weaver SC, Bellew LA, Rico-Hesse R. Phylogenetic analysis of alphaviruses in the Venezuelan equine encephalitis complex and identification of the source of epizootic viruses. Virology. 1992 Nov;191(1):282-90. doi: 10.1016/0042-6822(92)90190-z. PMID 1413507
- [Background] Young NA, Johnson KM. Antigenic variants of Venezuelan equine encephalitis virus: their geographic distribution and epidemiologic significance. Am J Epidemiol. 1969 Mar;89(3):286-307. doi: 10.1093/oxfordjournals.aje.a120942. No abstract available. PMID 5773424
- [Result] Martin DH, Eddy GA, Sudia WD, Reeves WC, Newhouse VF, Johnson KM. An epidemiologic study of Venezuelan equine encephalomyelitis in Costa Rica, 1970. Am J Epidemiol. 1972 Jun;95(6):565-78. doi: 10.1093/oxfordjournals.aje.a121426. No abstract available. PMID 5063895